CLINICAL TRIAL: NCT00552305
Title: An Open-label Extension Trial to Determine Tolerability and Efficacy of Long-term Oral SPM 927 as Adjunctive Therapy in Patients With Partial Seizures
Brief Title: To Determine Tolerability and Efficacy of Long-term Oral Lacosamide in Patients With Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0615
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Partial Epilepsies
MeSH Terms: conditions — Epilepsies, Partial | interventions — Lacosamide

ARMS (1):
- Lacosamide (Experimental): 50mg and 100mg tablets up to 800 mg/day as twice a day (BID) dosing
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — 50mg and 100mg tablets up to 800 mg/day as twice a day (BID) dosing throughout the trial
  Other Names: Vimpat

SUMMARY:
The purpose of this trial is to determine whether lacosamide is safe and effective for long-term use in patients with partial-seizures from epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Completion of parent clinical trial for treatment of partial seizures.

Exclusion Criteria:

* Receiving any study drug or experimental device other than lacosamide.
* Meets withdrawal criteria for parent trial or experiencing ongoing serious adverse event.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2001-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (59):
- United States (43):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Englewood, Colorado
  - Gainesville, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Ponte Vedra Beach, Florida
  - Chicago, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Wichita, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Frederick, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Saint Paul, Minnesota
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Somerset, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Irving, Texas
  - Lubbock, Texas
  - Wichita Falls, Texas
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
- Germany (4):
  - Bonn
  - Erlangen
  - Kehl Kork
  - Schwalmstedt-Treysa
- Hungary (2):
  - Budapest
  - Zalaegerszeg
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poznan, Poland
- Sweden (2):
  - Gothenburg
  - Stockholm
- Switzerland (2):
  - Bern/Biel
  - Zurich
- United Kingdom (3):
  - Bucks/London
  - Glasgow
  - Liverpool

REFERENCES:
- [Derived] Rosenfeld W, Fountain NB, Kaubrys G, Ben-Menachem E, McShea C, Isojarvi J, Doty P; SP615 Study Investigators. Safety and efficacy of adjunctive lacosamide among patients with partial-onset seizures in a long-term open-label extension trial of up to 8 years. Epilepsy Behav. 2014 Dec;41:164-70. doi: 10.1016/j.yebeh.2014.09.074. Epub 2014 Oct 27. PMID 25461210
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started in August of 2001 with recruitment occurring in the United States, Germany, Hungary, Lithuania, Poland, Sweden, Switzerland, and the United Kingdom. The study had last patient last visit in February of 2010.
Groups:
- Lacosamide: 50mg and 100mg tablets of lacosamide up to 800 mg/day as twice daily (BID) dosing throughout the trial (flexible dosing)
Period: Overall Study
Arm/Group | Lacosamide
Started | 370
Completed | 120
Not Completed | 250
Not completed — Adverse Event | 43
Not completed — Lack of Efficacy | 120
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 44
Not completed — Lack of efficacy/withdrew consent | 1
Not completed — Lack of efficacy (LoE)/adverse event | 3
Not completed — Adverse event (AE)/withdrew (WD) consent | 2
Not completed — Unsatisfactory compliance | 11
Not completed — Poor compliance/lost to follow-up | 1
Not completed — AE/Other: prohibited drug required | 1
Not completed — LoE/WD consent/Other: cannot make visits | 1
Not completed — Other: Site closed | 4
Not completed — Other: Personal problems | 1
Not completed — Other: Unable to attend visits | 1
Not completed — Other: Subject underwent surgery | 4
Not completed — Other: Subject became pregnant | 1
Not completed — Other: Health problems, not drug related | 1
Not completed — Other: Subject moved from area | 2
Not completed — Other: Subject incarcerated | 1
Not completed — Other: Subject went to rehab | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 370
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 364
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 178
Region of Enrollment [Number; unit: participants]
  United States | 248
  Hungary | 13
  Poland | 4
  Lithuania | 46
  Germany | 21
  United Kingdom | 12
  Switzerland | 2
  Sweden | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treat-Emergent Adverse Event (TEAE) During the Treatment Period (up to 8 Years)
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: During the Treatment Period (up to 8 years)
Population: Of the 370 subjects who entered the study, 370 are included in this summary based on the Safety Set (SS). SS population: number of subjects treated.
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 370
subjects | 343

2. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a Treatment-Emergent Adverse Event (TEAE) During the Treatment Period (up to 8 Years)
Description: as for outcome 1
Time Frame: During the Treatment Period (up to 8 years)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 370
subjects | 47

3. Primary Outcome: Number of Subjects Reporting at Least 1 Serious Adverse Event (SAE) During the Treatment Period (up to 8 Years)
Description: A serious adverse event is any untoward medical occurrences in a subject administered study treatment, whether or not the event is related to treatment, with at least one of the follow outcomes: death, life-threatening, initial inpatient hospitalization or prolongation of hospitalization, significant or persistent disability/incapacity, congenital anomaly/birth defect, or an important medical event that may jeopardize the subject and require a medical/surgical intervention.
Time Frame: During the Treatment Period (up to 8 years)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 370
subjects | 125

4. Secondary Outcome: Median Percentage Change From Baseline in 28-day Seizure Frequency During the Treatment Period (up to 8 Years)
Description: Median percentage change is the median value with respect to the percent change from Baseline across the population of subjects. Percentage change is calculated as 100 times the difference of the seizure frequency for the treatment period and the Baseline seizure frequency divided by the baseline seizure frequency.
  Negative changes from Baseline indicate an improvement (i.e., a reduction) in 28-day seizure frequency.
Time Frame: Baseline, End of Treatment Period (up to 8 years)
Population: Of the 370 subjects who were enrolled/treated in the study, 369 are included in this summary based on the Full Analysis Set (FAS). FAS population: number of subjects treated with at least 1 post-baseline seizure diary day with available data during the SP615 study.
Measure: Median (Full Range); unit: percentage change
Arm/Group | Lacosamide
Number analyzed (Participants) | 369
percentage change | -50.8 [-100.0 to 408.9]

5. Secondary Outcome: Percentage of at Least 50% Responders During the Treatment Period (up to 8 Years)
Description: At least 50 percent response is based on the percentage reduction in 28-day seizure frequency during the Treatment Period of the open-label extension relative to the Baseline Phase of the prior study. This endpoint reflects the percentage of subjects with at least 50% reduction (ie, at least 50% change) in 28-day partial onset seizure frequency
Time Frame: Treatment Period (up to 8 years)
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 369
percentage of subjects | 51.2

ADVERSE EVENTS:
Time Frame: The adverse event summaries are based on data collected during the 8 years of the study for all 370 patients
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 125/370
Other Adverse Events (participants affected / at risk) | 307/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=370)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 3 (3)
ANGINA PECTORIS (Cardiac disorders) | 3 (3)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (3)
COLITIS (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (2)
ENTEROCELE (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 5 (6)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (4)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
IRRITABILITY (General disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 3 (3)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
INJURY (Injury, poisoning and procedural complications) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 2 (2)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 2 (2)
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 (1)
TREATMENT NONCOMPLIANCE (Injury, poisoning and procedural complications) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (2)
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1)
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 1 (1)
ELECTROENCEPHALOGRAM (Investigations) | 4 (4)
ELECTROCARDIOGRAM QRS COMPLEX PROLONGED (Investigations) | 2 (2)
BIOPSY (Investigations) | 1 (1)
INVESTIGATION (Investigations) | 1 (1)
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 1 (1)
SINGLE PHOTON EMISSION COMPUTERISED TOMOGRAM (Investigations) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1)
ELECTROCARDIOGRAM CHANGE (Investigations) | 1 (1)
HEART RATE INCREASED (Investigations) | 1 (1)
URINARY CASTS (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (3)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 3 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CONVULSION (Nervous system disorders) | 23 (26)
STATUS EPILEPTICUS (Nervous system disorders) | 7 (7)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 (5)
HEADACHE (Nervous system disorders) | 3 (3)
HEMIPARESIS (Nervous system disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2)
GRAND MAL CONVULSION (Nervous system disorders) | 2 (2)
CEREBRAL INFARCTION (Nervous system disorders) | 2 (2)
EPILEPSY (Nervous system disorders) | 2 (2)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1)
MYASTHENIA GRAVIS CRISIS (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
COORDINATION ABNORMAL (Nervous system disorders) | 1 (1)
BALANCE DISORDER (Nervous system disorders) | 1 (2)
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 1 (1)
OPTIC NEURITIS RETROBULBAR (Nervous system disorders) | 1 (1)
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 1 (1)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 3 (3)
MAJOR DEPRESSION (Psychiatric disorders) | 2 (2)
AGGRESSION (Psychiatric disorders) | 2 (2)
SUICIDAL IDEATION (Psychiatric disorders) | 2 (2)
EPILEPTIC PSYCHOSIS (Psychiatric disorders) | 1 (2)
HALLUCINATION (Psychiatric disorders) | 1 (1)
PARANOIA (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (2)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1)
NIGHTMARE (Psychiatric disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (8)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 2 (2)
THERAPY REGIMEN CHANGED (Surgical and medical procedures) | 1 (1)
BRAIN OPERATION (Surgical and medical procedures) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1)
SURGERY (Surgical and medical procedures) | 1 (1)
BRAIN LOBECTOMY (Surgical and medical procedures) | 1 (1)
STENT PLACEMENT (Surgical and medical procedures) | 1 (1)
VAGAL NERVE STIMULATOR REMOVAL (Surgical and medical procedures) | 1 (1)
NASAL SEPTAL OPERATION (Surgical and medical procedures) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=370)
DIPLOPIA (Eye disorders) | 63 (92)
VISION BLURRED (Eye disorders) | 47 (60)
NAUSEA (Gastrointestinal disorders) | 64 (89)
VOMITING (Gastrointestinal disorders) | 49 (71)
DIARRHOEA (Gastrointestinal disorders) | 29 (40)
CONSTIPATION (Gastrointestinal disorders) | 20 (21)
FATIGUE (General disorders) | 61 (77)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 61 (108)
NASOPHARYNGITIS (Infections and infestations) | 60 (111)
SINUSITIS (Infections and infestations) | 43 (62)
INFLUENZA (Infections and infestations) | 32 (42)
URINARY TRACT INFECTION (Infections and infestations) | 31 (48)
BRONCHITIS (Infections and infestations) | 28 (34)
CONTUSION (Injury, poisoning and procedural complications) | 57 (129)
SKIN LACERATION (Injury, poisoning and procedural complications) | 50 (117)
EXCORIATION (Injury, poisoning and procedural complications) | 27 (50)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 19 (23)
WEIGHT INCREASED (Investigations) | 21 (22)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 43 (63)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 33 (49)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 31 (42)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 21 (30)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 20 (24)
DIZZINESS (Nervous system disorders) | 147 (254)
HEADACHE (Nervous system disorders) | 77 (145)
COORDINATION ABNORMAL (Nervous system disorders) | 53 (69)
SOMNOLENCE (Nervous system disorders) | 41 (50)
TREMOR (Nervous system disorders) | 39 (55)
MEMORY IMPAIRMENT (Nervous system disorders) | 27 (29)
CONVULSION (Nervous system disorders) | 27 (32)
BALANCE DISORDER (Nervous system disorders) | 26 (34)
NYSTAGMUS (Nervous system disorders) | 24 (28)
HYPOAESTHESIA (Nervous system disorders) | 20 (26)
INSOMNIA (Psychiatric disorders) | 33 (35)
DEPRESSION (Psychiatric disorders) | 33 (36)
ANXIETY (Psychiatric disorders) | 19 (20)
COUGH (Respiratory, thoracic and mediastinal disorders) | 29 (33)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 26 (34)
RASH (Skin and subcutaneous tissue disorders) | 28 (33)
HYPERTENSION (Vascular disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.